CLINICAL TRIAL: NCT06631118
Title: Pericapsular Nerve Group (PENG) Block Versus Low Dose Propofol to Achieve Painless Sitting Position Before Spinal Anesthesia in Patients With Hip Fractures
Brief Title: Pericapsular Nerve Block Versus Propofol During Hip Fractures Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwa Emam, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU R 130/2024
Record Dates: First submitted 2024-10-07; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Difference in Reduction in Visual Analogue Score at 30 Minutes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group (A ) : will receive ultrasound guided pericapsular nerve group block (PENG) followed by spinal anesthesia.
  Interventions: Procedure: pericapsular nerve group block for group A,low dose intravenous Propofol [0.7mg/kg] over 30 seconds for group B
- Group B (Active Comparator): Group B will receive low dose intravenous Propofol [0.7mg/kg] over 30 seconds followed by spinal anesthesia and so far, this is the most common and standard technique to achieve sitting position during spinal anesthesia for patients with hip fractures.
  Interventions: Procedure: pericapsular nerve group block for group A,low dose intravenous Propofol [0.7mg/kg] over 30 seconds for group B

INTERVENTIONS:
Procedure: pericapsular nerve group block for group A,low dose intravenous Propofol [0.7mg/kg] over 30 seconds for group B — Patients in group A will receive ultrasound guided pericapsular nerve group block (PENG) while patients in group B will receive low dose intravenous Propofol0.7mg/kg] over 30 seconds followed by spinal anesthesia in both groups

SUMMARY:
The study will compare the efficacy of Pericapsular nerve group block (PENG) versus low dose Propofol for the achievement of painless sitting position before spinal anesthesia in patients undergoing repair of Hip fractures.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the age group ranging 40-70, both genders, belonging to physical status American Society of Anaesthesiologists (ASA) I and II

Exclusion Criteria:

* Patients with old fractures (more than 7 days), polytrauma, bleeding disorders or coagulopathy, local site infection, difficulty expressing pain scores such as hearing disability, mentally challenged, dementia or psychiatric illness and who refused to take part

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-21 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
The difference in VAS scale | 30 min after giving propofol and the PENG block.
  The primary outcome will be difference in median reduction in VAS-D .

IPD SHARING:
Plan to Share IPD: Yes
Study protocol